CLINICAL TRIAL: NCT03666507
Title: Vegetative Monitoring During Brainstem-associated Surgery
Status: Completed | Type: Observational
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Other Study IDs: ANSTue
Record Dates: First submitted 2018-08-30; First posted 2018-09-11 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2021-04

CONDITIONS: Brain Tumor, Recurrent; Vestibular Schwannoma; Brainstem Neoplasm; Brainstem Glioma
MeSH Terms: conditions — Brain Neoplasms; Neuroma, Acoustic; Brain Stem Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Brain stem associated tumors: Brain stem associated tumors
  Interventions: Procedure: Intraoperative Monitoring during resection of brain tumor
- Tumors without brain stem assocation: Tumors without brain stem assocation
  Interventions: Procedure: Intraoperative Monitoring during resection of brain tumor

INTERVENTIONS:
Procedure: Intraoperative Monitoring during resection of brain tumor — Intraoperative Monitoring during resection of brain tumor

SUMMARY:
Intraoperative Monitoring of Heart rate variability, Blood pressure variability, Baroreceptorsensivity etc.

ELIGIBILITY:
Inclusion Criteria:

* age 0-99
* brain tumor

Exclusion Criteria:

* no consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Brain tumor patients
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2018-08-28 (Actual); Primary Completion 2020-08-28 (Actual); Study Completion 2021-03-28 (Actual)

PRIMARY OUTCOMES:
Heart rate variability (HRV) | intraoperatively
  Comparison of HRV in the 2 groups (brain stem-associated vs. non associated surgery)

SECONDARY OUTCOMES:
Rate of cardiovascular complications | intraoperatively
  Comparison of no. of cardiovascular complications (cardiac arrest, sudden tachy/bradyarryhthmia, hyper/hypotension, trigeminocardiac reflex) in the 2 groups

CONTACTS AND LOCATIONS:
Overall Officials: Martin U Schuhmann, Prof, Principal Investigator — University Hospital Tuebingen
Locations (1):
- Department of Neurosurgery, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: No